CLINICAL TRIAL: NCT01874535
Title: The Rates of Complete Symptom Relief,Prevetion of Symptom Relapse and Maintenance of Esophagitis Healing for 4-week Versus 8-week Esomeprazole Therapy Among Los Angeles Grades A and B Erosive Esophagitis
Brief Title: Rate of Complete Symptom Relief, Prevention of Symptom Relapse: Grades A and B Esophagitis of Esomeprazole Therapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Wei-Chen Tai M.D., Attending physician, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GERD A and B
Record Dates: First submitted 2012-11-04; First posted 2013-06-11 (Estimated); Results first posted 2018-09-04 (Actual); Last update posted 2018-09-04 (Actual); Status verified 2017-06

CONDITIONS: Erosive Esophagitis
MeSH Terms: interventions — Esomeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- GERD Los Angeles A and B-4 week group (Active Comparator): Patients with Los Angeles A and B esophagitis prescribed with esomeprazole (40 mg)daily- 4 week group
  Interventions: Drug: Esomeprazole 40 mg
- GERD Los Angeles A and B-8-week group (Active Comparator): Patients with Los Angeles A and B esophagitis prescribed with esomeprazole (40 mg)daily- 8 week group
  Interventions: Drug: Esomeprazole 40 mg

INTERVENTIONS:
Drug: Esomeprazole 40 mg — Comparison of 4-weeks and 8-weeks initial treatment duration of esomeprazole 40 mg per day on the rate of symptom relapse and sustained healing of esophagitis in patients with symptomatic erosive esophagitis
  Other Names: Nexium 40mg

SUMMARY:
To investigate the impact of initial treatment duration (4-week versus 8-week)of Esomeprazole (40mg) on the rate of symptom relapse and sustained healing of esophagitis in patients with symptomatic erosive esophagitis

DETAILED DESCRIPTION:
Patients:

Patients between the ages of 15 and 80 years with clinical symptoms of acid regurgitation, heart burn, or feeling of acidity in the stomach, who have Los Angeles Grade A and B erosive esophagitis proven by endoscopy are recruited. Criteria for exclusions include (1) coexistence of peptic ulcer or gastrointestinal malignancies, (2) pregnancy, (3) coexistence of serious concomitant illness (for example, decompensated liver cirrhosis and uremia), (4) previous gastric surgery, (5) allergy to esomeprazole, (6) symptom score of a validated questionnaire (Chinese GERDQ) less than 12, and (7) equivocal endoscopic diagnosis of Los Angeles Grade A and B erosive esophagitis.

Outcome parameters:

The main outcome measures

1. Rate of complete symptom relief (CSR) at the end of initial treatment phase
2. rate of symptom relapse within 12 weeks after stopping initial therapy

ELIGIBILITY:
Inclusion Criteria:

* patients between the ages of 15 and 80 years
* with clinical symptoms of acid regurgitation, heart burn, or feeling of acidity in the stomach,
* who have Los Angeles Grade A and B erosive esophagitis proven by endoscopy are recruited.

Exclusion Criteria:

1. coexistence of peptic ulcer or gastrointestinal malignancies,
2. pregnancy,
3. coexistence of serious concomitant illness (for example, decompensated liver cirrhosis and uremia),
4. previous gastric surgery,
5. allergy to esomeprazole,
6. symptom score of a validated questionnaire (Chinese GERDQ) less than 12, and
7. equivocal endoscopic diagnosis of Los Angeles Grade A and B erosive esophagitis.

Ages: 15 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 408 (Actual)
Dates: Start 2010-06; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Seng-Kee Chuah, M.D, Study Chair — Kaohsiung Chang Gung Memorial Hospital,Taiwan
Locations (1):
- Seng-Kee Chuah, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
The data will be shared in July 2017

REFERENCES:
- [Derived] Hsu PI, Lu CL, Wu DC, Kuo CH, Kao SS, Chang CC, Tai WC, Lai KH, Chen WC, Wang HM, Cheng JS, Tsai TJ, Chuah SK. Eight weeks of esomeprazole therapy reduces symptom relapse, compared with 4 weeks, in patients with Los Angeles grade A or B erosive esophagitis. Clin Gastroenterol Hepatol. 2015 May;13(5):859-66.e1. doi: 10.1016/j.cgh.2014.09.033. Epub 2014 Sep 20. PMID 25245625

RESULTS

PARTICIPANT FLOW:
Groups:
- 4-week Group: Patients with Los Angeles A and B esophagitis prescribed with esomeprazole (40 mg)daily
  Esomeprazole 40 mg: Comparison of 4-weeks initial treatment duration of esomeprazole 40 mg per day on the rate of symptom relapse and sustained healing of esophagitis in patients with symptomatic erosive esophagitis
- 8-week Group: Patients with Los Angeles A and B esophagitis prescribed with esomeprazole (40 mg)daily
  Esomeprazole 40 mg: Comparison of 8-weeks initial treatment duration of esomeprazole 40 mg per day on the rate of symptom relapse and sustained healing of esophagitis in patients with symptomatic erosive esophagitis
Period: Overall Study
Arm/Group | 4-week Group | 8-week Group
Started | 207 | 201
Completed | 152 | 157
Not Completed | 55 | 44
Not completed — Lost to Follow-up | 10 | 9
Not completed — incomplete symptom resolution | 45 | 35

BASELINE CHARACTERISTICS:
Population: Baseline characteristics of the enrolled patients
Groups:
- Total: Total of all reporting groups
Arm/Group | 4-week Group | 8-week Group | Total
Number analyzed (Participants) | 207 | 201 | 408
Age, Continuous [Mean (Standard Deviation); unit: years]
  age | 51.1 (12.8) | 51.1 (12.8) | 51.1 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  sex: Female | 87 | 77 | 164
  sex: Male | 120 | 124 | 244
Region of Enrollment [Count of Participants; unit: Participants]
  Taiwan | 207 | 201 | 408

OUTCOME MEASURES:

1. Primary Outcome: The Rates of Complete Symptom Relief
Description: Rate of complete symptom relief (CSR) at the end of initial treatment phase
Time Frame: at the 20 weeks after the end of initial treatment.
Measure: Number; unit: participants
Groups:
- 4 Week Group: Patients with Los Angeles A and B esophagitis prescribed with esomeprazole (40 mg)daily
  Esomeprazole 40 mg: Comparison of 4-weeks weeks initial treatment duration of esomeprazole 40 mg per day on the rate of symptom relapse and sustained healing of esophagitis in patients with symptomatic erosive esophagitis
- 8 Week Group: Patients with Los Angeles A and B esophagitis prescribed with esomeprazole (40 mg)daily
  Esomeprazole 40 mg: Comparison of 8-weeks initial treatment duration of esomeprazole 40 mg per day on the rate of symptom relapse and sustained healing of esophagitis in patients with symptomatic erosive esophagitis
Arm/Group | 4 Week Group | 8 Week Group
Number analyzed (Participants) | 207 | 201
participants | 152 | 157
Statistical Analysis 1: Comparison: 4 Week Group vs 8 Week Group; Test type: Superiority or Other; p < 0.05, Chi-squared; Hazard Ratio (HR) = 0.009

ADVERSE EVENTS:
Time Frame: 20 weeks
Groups:
- 4 Week Group: Patients with Los Angeles A and B esophagitis prescribed with esomeprazole (40 mg)daily
  Esomeprazole 40 mg: Comparison of 4-weeks initial treatment duration of esomeprazole 40 mg per day on the rate of symptom relapse and sustained healing of esophagitis in patients with symptomatic erosive esophagitis
Arm/Group | 4 Week Group | 8 Week Group
All-Cause Mortality (participants affected / at risk) | 0/207 | 0/201
Serious Adverse Events (participants affected / at risk) | 0/207 | 0/201
Other Adverse Events (participants affected / at risk) | 0/207 | 0/201

LIMITATIONS AND CAVEATS:
The trial was performed in a single country

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No